CLINICAL TRIAL: NCT02986230
Title: Implementing Cancer Prevention Using Patient-Provider Clinical Decision Support
Brief Title: Cancer Prevention Clinical Decision Support
Acronym: CP-CDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-010
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2022-02

CONDITIONS: Cancer Prevention
Keywords: Cancer prevention; Clinical Decision Support; Rural Health; Shared Decision Making

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CP-CDS (Experimental): The CP-CDS group will receive a point of care clinical decision support tool called cancer prevention wizard (CP Wizard) that is integrated into the EHR. The CP Wizard provides evidenced- based recommendations to the provider and patient related to overdue cancer prevention screening services.
  Interventions: Other: CP-CDS
- CP-CDS + SDMT (Experimental): The CP-CDS + SDMT group will receive a point of care clinical decision support tool called cancer prevention wizard (CP Wizard) that is integrated into the EHR. The CP Wizard provides evidenced- based recommendations to the provider and patient related to overdue cancer prevention screening services. The CP-CDS + SDMT arm also provides shared decision making tools to patient and provider at the time of the visit.
  Interventions: Other: CP-CDS
- Usual Care (No Intervention): The usual care group will have no access to the CP-CDS, or the CP-CDS + SDMT.

INTERVENTIONS:
Other: CP-CDS — The cancer prevention wizard is a point of care clinical decision support system designed to identify patients that are due for preventative cancer services and provides evidenced-based recommendations to the patient and provider.
  Other Names: Cancer Prevention Wizard
  Arms: CP-CDS; CP-CDS + SDMT

SUMMARY:
The objective of this project is to implement and evaluate the effectiveness of a sophisticated Web-based, electronic health record (EHR)-linked clinical decision support (CDS) system designed to improve primary and secondary cancer preventive care.

This project will engage a rural population with substantial healthcare disparities and gaps in the receipt of primary and secondary cancer prevention. Results will advance dissemination and implementation research methods that can reduce health disparities and improve healthcare for millions in medically under-served areas.

DETAILED DESCRIPTION:
The objective of this project is to implement and evaluate the effectiveness of a sophisticated Web-based, electronic health record (EHR)-linked clinical decision support (CDS) system designed to improve primary and secondary cancer preventive care. To achieve this objective, EHR data is sent to evidence-based cancer prevention algorithms, housed on a secure Web site. The algorithms: (a) identify at the point of care all eligible patients not up to date on their cancer prevention interventions; and (b) present to both patient and primary care provider (PCP), appropriate evidence-based primary cancer prevention interventions and cancer screening options at the point of care. The cancer prevention (CP)-CDS will focus on breast cancer screening in women aged 50-74, colorectal cancer screening for both sexes aged 50-75, cervical cancer screening for women aged 21-65, human papilloma virus (HPV) vaccination for both sexes aged 11-26, and referrals for weight management and smoking cessation in all adults aged 18 and older. Effectiveness is assessed by cluster-randomizing 30 primary care clinics with roughly 285 PCPs and 153,000 study-eligible patients into one of three experimental conditions: Group 1: CP-CDS intervention in which the decision support is printed for the PCP and patient, designed to engage patients in discussions about appropriate cancer prevention strategies. Group 2: CP-CDS + shared decision making tools (SDMT) intervention in which the CP-CDS is printed along with additional shared decision making tools. Group 3: clinics provide usual care (UC) with no intervention-related activity related to cancer prevention.

With 10 clinics, 95 PCPs, and 51,000 potentially eligible patients per study arm, this study will formally test the hypothesis that Groups 1 and 2 are superior to Group 3 over an 12-month follow-up period with respect to: (a) significantly higher rates of appropriate screening for breast, cervix, and colorectal cancer, as defined by the United States Preventive Services Task Force; and (b) significantly higher rates of human papillomavirus (HPV) vaccination in males and females aged 11-26 years. Secondary analysis will evaluate the impact of the intervention on lung cancer screening. The investigators further posit that Groups 1 and 2 will have higher short-term health care costs but better long-term cost-effectiveness than Group 3. The Consolidated Framework for Implementation Research (CFIR) and Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) conceptual frameworks will be used to guide implementation planning, organization, conduct, and impact evaluation of the intervention in a large rural healthcare system.

This project will engage a rural population with substantial healthcare disparities and gaps in the receipt of primary and secondary cancer prevention. Results will advance dissemination and implementation research methods that can reduce health disparities and improve healthcare for millions in medically under-served areas.

ELIGIBILITY:
Inclusion Criteria:

* meet above age criteria
* pcp practice at randomized clinic

Exclusion Criteria:

* current or past cancer diagnosis (excludes nonmelanoma skin cancer)
* hospice care or cancer chemotherapy
* Alzheimer's disease codes
* major cardiovascular event in 12 months prior to index date

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35953 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Elliott, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- Essentia Health, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliott TE, O'Connor PJ, Asche SE, Saman DM, Dehmer SP, Ekstrom HL, Allen CI, Bianco JA, Chrenka EA, Freitag LA, Harry ML, Truitt AR, Sperl-Hillen JM. Design and rationale of an intervention to improve cancer prevention using clinical decision support and shared decision making: A clinic-randomized trial. Contemp Clin Trials. 2021 Mar;102:106271. doi: 10.1016/j.cct.2021.106271. Epub 2021 Jan 24. PMID 33503497
- [Background] Harry ML, Chrenka EA, Freitag LA, Saman DM, Allen CI, Asche SE, Truitt AR, Ekstrom HL, O'Connor PJ, Sperl-Hillen JAM, Ziegenfuss JY, Elliott TE. Primary care clinicians' opinions before and after implementation of cancer screening and prevention clinical decision support in a clinic cluster-randomized control trial: a survey research study. BMC Health Serv Res. 2022 Jan 6;22(1):38. doi: 10.1186/s12913-021-07421-0. PMID 34991570
- [Background] Saman DM, Harry ML, Freitag LA, Allen CI, O'Connor PJ, Sperl-Hillen JM, Bianco JA, Truitt AR, Ekstrom HL, Elliott TE. Patient Perceptions of Using Clinical Decision Support for Cancer Screening and Prevention: "I wouldn't have thought about getting screened without it.". J Patient Cent Res Rev. 2021 Oct 18;8(4):297-306. doi: 10.17294/2330-0698.1863. eCollection 2021 Fall. PMID 34722797
- [Background] Saman DM, Chrenka EA, Harry ML, Allen CI, Freitag LA, Asche SE, Truitt AR, Ekstrom HL, O'Connor PJ, Sperl-Hillen JM, Ziegenfuss JY, Elliott TE. The impact of personalized clinical decision support on primary care patients' views of cancer prevention and screening: a cross-sectional survey. BMC Health Serv Res. 2021 Jun 21;21(1):592. doi: 10.1186/s12913-021-06551-9. PMID 34154588
- [Background] Harry ML, Saman DM, Truitt AR, Allen CI, Walton KM, O'Connor PJ, Ekstrom HL, Sperl-Hillen JM, Bianco JA, Elliott TE. Pre-implementation adaptation of primary care cancer prevention clinical decision support in a predominantly rural healthcare system. BMC Med Inform Decis Mak. 2020 Jun 23;20(1):117. doi: 10.1186/s12911-020-01136-8. PMID 32576202
- [Background] Saman DM, Walton KM, Harry ML, Asche SE, Truitt AR, Henzler-Buckingham HA, Allen CI, Ekstrom HL, O'Connor PJ, Sperl-Hillen JM, Ziegenfuss JY, Bianco JA, Elliott TE. Understanding primary care providers' perceptions of cancer prevention and screening in a predominantly rural healthcare system in the upper Midwest. BMC Health Serv Res. 2019 Dec 30;19(1):1019. doi: 10.1186/s12913-019-4872-9. PMID 31888630
- [Background] Harry ML, Truitt AR, Saman DM, Henzler-Buckingham HA, Allen CI, Walton KM, Ekstrom HL, O'Connor PJ, Sperl-Hillen JM, Bianco JA, Elliott TE. Barriers and facilitators to implementing cancer prevention clinical decision support in primary care: a qualitative study. BMC Health Serv Res. 2019 Jul 31;19(1):534. doi: 10.1186/s12913-019-4326-4. PMID 31366355
- [Background] Harry ML, Asche SE, Freitag LA, Sperl-Hillen JM, Saman DM, Ekstrom HL, Chrenka EA, Truitt AR, Allen CI, O'Connor PJ, Dehmer SP, Bianco JA, Elliott TE. Human Papillomavirus vaccination clinical decision support for young adults in an upper midwestern healthcare system: a clinic cluster-randomized control trial. Hum Vaccin Immunother. 2022 Dec 31;18(1):2040933. doi: 10.1080/21645515.2022.2040933. Epub 2022 Mar 18. PMID 35302909
- [Background] Elliott TE, Asche SE, O'Connor PJ, Dehmer SP, Ekstrom HL, Truitt AR, Chrenka EA, Harry ML, Saman DM, Allen CI, Bianco JA, Freitag LA, Sperl-Hillen JM. Clinical Decision Support with or without Shared Decision Making to Improve Preventive Cancer Care: A Cluster-Randomized Trial. Med Decis Making. 2022 Aug;42(6):808-821. doi: 10.1177/0272989X221082083. Epub 2022 Feb 25. PMID 35209775

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were accrued if they were not up to date on breast, cervical, or colorectal cancer screening, or not up to date on HPV vaccine at the index visit. Eligibility was determined using automated algorithms.
Pre-assignment Details: Cluster randomization of the 34 primary care clinics was done to minimize contamination. Pre-randomization balance factors included: 1) clinic urbanicity, and 2) percentage of women at each clinic up to date on breast cancer screening. The first concealed randomization scheme meeting balance criteria was selected. 35953 participants were allocated to one of three groups (i.e. Started). The number Completed reflects the number of subjects included in final analysis after exclusions and opt outs.
Units Other Than Participants: primary care clinics
Groups:
- CP-CDS + SDMT: The SDMT-focused group will receive the point of care clinical decision support tool called cancer prevention wizard (CP Wizard) that is integrated into the EHR. The CP Wizard provides evidenced- based recommendations to the provider and patient related to overdue cancer prevention screening services. The SDMT-focused arm also provides shared decision making tools to patient and provider at the time of the visit.
  CP-CDS: The cancer prevention wizard is a point of care clinical decision support system designed to identify patients that are due for preventative cancer services and provides evidenced-based recommendations to the patient and provider.
- Usual Care: Patients of providers practicing at clinics assigned to the usual care arm will have no access to the CP-CDS or CP-CDS + SDMTs.
Period: Overall Study
Arm/Group | CP-CDS | CP-CDS + SDMT | Usual Care
Started | 11402; 11 primary care clinics | 10138; 11 primary care clinics | 14413; 12 primary care clinics
Completed | 10122; 11 primary care clinics | 9034; 11 primary care clinics | 12960; 12 primary care clinics
Not Completed | 1280; 0 primary care clinics | 1104; 0 primary care clinics | 1453; 0 primary care clinics

BASELINE CHARACTERISTICS:
Population: Analysis population included patients not up to date on one or more composite screening for breast, cervical, or colorectal cancer, HPV vaccine, or lung cancer screening.
Groups:
- CP-CDS: Providers practicing in the PCP-focused group will receive a point of care clinical decision support tool called cancer prevention wizard (CP Wizard) that is integrated into the EHR. The CP Wizard provides evidenced- based recommendations to the provider and patient related to overdue cancer prevention screening services.
  CP-CDS: The cancer prevention wizard is a point of care clinical decision support system designed to identify patients that are due for preventative cancer services and provides evidenced-based recommendations to the patient and provider.
- CP-CDS + SDMT: Providers practicing in the SDMT-focused group will receive a point of care clinical decision support tool called cancer prevention wizard (CP Wizard) that is integrated into the EHR. The CP Wizard provides evidenced- based recommendations to the provider and patient related to overdue cancer prevention screening services. The SDMT-focused arm also provides shared decision making tools to patient and provider at the time of the visit.
  CP-CDS: The cancer prevention wizard is a point of care clinical decision support system designed to identify patients that are due for preventative cancer services and provides evidenced-based recommendations to the patient and provider.
- Usual Care: Providers practicing at clinics assigned to the usual care arm will have no access to the CP Wizard.
- Total: Total of all reporting groups
Arm/Group | CP-CDS | CP-CDS + SDMT | Usual Care | Total
Number analyzed (Participants) | 10122 | 9034 | 12960 | 32116
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (17.2) | 47.9 (17.5) | 47.7 (17.3) | 48.0 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6725 | 5870 | 8532 | 21127
  Male | 3397 | 3164 | 4428 | 10989
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 116 | 100 | 181 | 397
  Not Hispanic or Latino | 9917 | 8863 | 12670 | 31450
  Unknown or Not Reported | 89 | 71 | 109 | 269
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 261 | 169 | 155 | 585
  Asian | 74 | 65 | 72 | 211
  Native Hawaiian or Other Pacific Islander | 19 | 9 | 26 | 54
  Black or African American | 164 | 122 | 199 | 485
  White | 9459 | 8548 | 12343 | 30350
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 145 | 121 | 165 | 431

OUTCOME MEASURES:

1. Primary Outcome: Composite Cancer Screening Tests up to Date
Description: Participants up to date on composite endpoint of breast, cervical, and colorectal cancer screening at 1 year post index date.
Time Frame: 1 year post index date
Population: Analysis population included adult patients ages 21-75 who had a visit at a study clinic over the accrual period, and who were due for one or more breast, cervical, or colorectal cancer screening test.
Measure: Count of Participants; unit: Participants
Groups:
- CP-CDS: The PCP-focused group will receive a point of care clinical decision support tool called cancer prevention wizard (CP Wizard) that is integrated into the EHR. The CP Wizard provides evidenced- based recommendations to the provider and patient related to overdue cancer prevention screening services.
  CP-CDS: The cancer prevention wizard is a point of care clinical decision support system designed to identify patients that are due for preventative cancer services and provides evidenced-based recommendations to the patient and provider.
- CP-CDS + SDMT: The SDMT-focused group will receive a point of care clinical decision support tool called cancer prevention wizard (CP Wizard) that is integrated into the EHR. The CP Wizard provides evidenced- based recommendations to the provider and patient related to overdue cancer prevention screening services. The SDMT-focused arm also provides shared decision making tools to patient and provider at the time of the visit.
  CP-CDS: The cancer prevention wizard is a point of care clinical decision support system designed to identify patients that are due for preventative cancer services and provides evidenced-based recommendations to the patient and provider.
Arm/Group | CP-CDS | CP-CDS + SDMT | Usual Care
Number analyzed (Participants) | 7987 | 7105 | 10106
Participants | 3087 | 2590 | 3866
Statistical Analysis 1: Comparison: CP-CDS vs Usual Care; Generalized linear mixed models with logit link and binomial error distribution were used to test the effect of the intervention on the composite of cancer screening by 1 year post-index for breast, cervical, and colorectal cancer. The model included two primary contrasts: CP-CDS vs. UC and CP-CDS+SDMT vs. UC and included pre-specified covariates and variables used in the randomization process. Tests of the two contrasts were 2-sided with P-values < 0.025 considered statistically significant; Test type: Superiority; p = .025, Mixed Models Analysis — Tests of the two planned contrasts were 2-sided with P-values less than 0.025 considered statistically significant, and odds ratios for key study group contrasts report 97.5% confidence intervals; Denominator degrees of freedom for variables in the model take into account the cluster-randomized design; Odds Ratio (OR) = 1.07
Statistical Analysis 2: Comparison: CP-CDS + SDMT vs Usual Care; Generalized linear mixed models with a logit link and binomial error distribution were used to test the effect of the intervention on the composite of cancer screening by 1 year post-index date for breast, cervical, and colorectal cancer. Model included two primary contrasts: CP-CDS vs. UC and CP-CDS+SDMT vs. UC and included pre-specified covariates and variables used in randomization process. Tests of the planned contrasts were 2-sided with P-values < 0.025 considered statistically significant; Test type: Superiority; p = .025, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Denominator degrees of freedom for variables in the model take into account the cluster-randomized design; Odds Ratio (OR) = 0.91

2. Primary Outcome: HPV Vaccination up to Date
Description: Participants up to date on HPV vaccination at 1 year post index date.
Time Frame: 1 year post index date
Population: Young adults ages 18-26 with a visit at a study clinic during the accrual period, and not up to date on HPV vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | CP-CDS | CP-CDS + SDMT | Usual Care
Number analyzed (Participants) | 1511 | 1470 | 2073
Participants | 90 | 69 | 126
Statistical Analysis 1: Comparison: CP-CDS vs Usual Care; Generalized linear mixed models with a logit link and binomial error distribution were used to test the effect of the intervention on completion of the HPV vaccination series by 12 months post-index date. The model included two primary contrasts: CP-CDS vs. UC and CP-CDS+SDMT vs. UC and included pre-specified covariates and variables used in the randomization process. Tests of the two planned contrasts were 2-sided with P-values less than 0.025 considered statistically significant; Test type: Superiority; p = .025, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Denominator degrees of freedom for variables in the model take into account the cluster-randomized design; Odds Ratio (OR) = 1.04
Statistical Analysis 2: Comparison: CP-CDS + SDMT vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .025, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Denominator degrees of freedom for variables in the model take into account the cluster-randomized design; Odds Ratio (OR) = 0.71

3. Secondary Outcome: Lung Cancer Screening up to Date
Description: Participants up to date on lung cancer screening at 1 year post index date.
Time Frame: 1 year post index date
Population: Adult patients with a visit at a study clinic and not up to date for lung cancer screening at index date.
Measure: Count of Participants; unit: Participants
Arm/Group | CP-CDS | CP-CDS + SDMT | Usual Care
Number analyzed (Participants) | 624 | 459 | 781
Participants | 200 | 104 | 198
Statistical Analysis 1: Comparison: CP-CDS vs Usual Care; Generalized linear mixed models with a logit link and binomial error distribution were used to test the effect of the intervention on completion of lung cancer screening by 12 months post-index date. The model included two primary contrasts: CP-CDS vs. UC and CP-CDS+SDMT vs. UC and included pre-specified covariates and variables used in the randomization process. Tests of the two planned contrasts were 2-sided with P-values less than 0.025 considered statistically significant; Test type: Superiority; p = .025, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Denominator degrees of freedom for variables in the model take into account the cluster-randomized design; Odds Ratio (OR) = 1.55
Statistical Analysis 2: Comparison: CP-CDS + SDMT vs Usual Care; Generalized linear mixed models with a logit link and binomial error distribution were used to test the intervention effect on the completion of lung cancer screening by 12 months post-index. The model included two primary contrasts: CP-CDS vs. UC and CP-CDS+SDMT vs. UC and included pre-specified covariates and variables used in the randomization process. Tests of the two planned contrasts were 2-sided with P-values less than 0.025 considered statistically significant; Test type: Superiority; p = .025, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Denominator degrees of freedom for variables in the model take into account the cluster-randomized design; Odds Ratio (OR) = 1.02

ADVERSE EVENTS:
Time Frame: Actual compared to expected accrual was reported at 6 months, 12 months, and 15 months.
Description: This is a minimal risk study designed to improve cancer screening rates. Feedback from providers on the CDS tool was monitored and printing rates for the CDS interface were monitored.
Groups:
- CP-CDS: Providers in the PCP-focused group will receive a point of care clinical decision support tool called cancer prevention wizard (CP Wizard) that is integrated into the EHR. The CP Wizard provides evidenced- based recommendations to the provider and patient related to overdue cancer prevention screening services.
  CP-CDS: The cancer prevention wizard is a point of care clinical decision support system designed to identify patients that are due for preventative cancer services and provides evidenced-based recommendations to the patient and provider.
- CP-CDS + SDMT: Providers in the SDMT-focused group will receive a point of care clinical decision support tool called cancer prevention wizard (CP Wizard) that is integrated into the EHR. The CP Wizard provides evidenced- based recommendations to the provider and patient related to overdue cancer prevention screening services. The SDMT-focused arm also provides shared decision making tools to patient and provider at the time of the visit.
  CP-CDS: The cancer prevention wizard is a point of care clinical decision support system designed to identify patients that are due for preventative cancer services and provides evidenced-based recommendations to the patient and provider.
Arm/Group | CP-CDS | CP-CDS + SDMT | Usual Care
All-Cause Mortality (participants affected / at risk) | 22/10122 | 15/9034 | 26/12960
Serious Adverse Events (participants affected / at risk) | 0/10122 | 0/9034 | 0/12960
Other Adverse Events (participants affected / at risk) | 0/10122 | 0/9034 | 0/12960

LIMITATIONS AND CAVEATS:
The study was conducted at one relatively high-performing predominantly rural healthcare system, and generalizability of results to other care systems or patient populations is uncertain. The intervention was delivered during clinic encounters with primary care providers; the impact of the clinical decision support delivered in other clinical venues or directly to patients using mobile health technologies may be greater or less than what we observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT02986230/Prot_SAP_000.pdf